CLINICAL TRIAL: NCT07289594
Title: The Impact of Psychosocial Support Web-based Toolkit on Psychological Immunity, Self-care Behaviors, and Job Performance Among ECD Frontliners in Lebanon
Brief Title: Impact of Psychosocial Support Web-Based Toolkit
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arab Resource Collective (Other)
Collaborators: Modern University for Business and Science (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MU-20250122-53
Record Dates: First submitted 2025-11-19; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Mental Health; Self Care; Performance Enhancement
Keywords: Mental Health; Early Childhood Development (ECD); Psychological Immunity; Cognitive Emotional Regulation; Self Care Behaviors; Job Performance; Web-based Toolkit; Psychosocial Support
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MHPSS Web-Based Toolkit Intervention (Experimental): Participants will receive a web-based psychosocial support toolkit designed to enhance psychological immunity, self-care behaviors, and job performance among Early Childhood Development (ECD) frontliners in Lebanon. This Toolkit consists of (10) online sessions delivered in an interactive digital way.
  Interventions: Behavioral: MHPSS Web-Based Toolkit

INTERVENTIONS:
Behavioral: MHPSS Web-Based Toolkit — An intervention that is delivered through an online toolkit that aims to improve psychological immunity, self-care behaviors, and job performance among ECD frontliners.
  Other Names: Impact of Online Toolkit; Web-Based Psychosocial Support Toolkit

SUMMARY:
At times of crisis, early childhood development (ECD) workers, and schools/centers play an important role in the lives of children in the early childhood stage (less than 8 years old) and their parents; they are intended to act as the "great equalizer", offering not only curriculum teaching, but also additional social-emotional learning and educational opportunities for vulnerable children who are more likely to suffer in such situations.

CD teachers, despite this responsibility, often lack tools and methods to promote their well-being, and to cope with vulnerable children and difficult situations. They are also rarely recognized as members of a workforce with specialized knowledge or competencies, and they hardly receive the support needed to uphold this great responsibility to young children, their families, and society.

DETAILED DESCRIPTION:
ECD frontliners working in the field might face many challenges, stories, and situations that affect their mental health and could cause them distress and complications. Hence, these negative consequences could affect their ability to perform their jobs and provide the services they usually provide with the same quality. It might also affect their ability to respond to the children's emotional and social needs.

It was reported that ECD frontliners, such as teachers and instructors, have the highest levels of psychological symptoms, such as anxiety, in addition to high levels of stress and low levels of well-being. Findings indicate that ECD frontliners who already struggle with poor well-being and poor working conditions will suffer more from emotional and physical burdens while working with children, especially vulnerable children.

A study made by Kwon et al. (2019) found a positive significant relationship between the depressive symptoms of ECD teachers, the quality of emotional and behavioral support ECD teachers provide, and the behavioral problems of their students. According to this study, teachers with depressive symptoms are less likely to provide positive emotional and behavioral support to children since these symptoms may limit their ability to provide warm care and nurturing environments. Moreover, due to their psychological stress, teachers may exhibit negative moods, poor behavioral modeling, and poor self-regulation, which the children may respond to and learn from. Hence, providing sensitive-responsive interactions and nurturing environments for children in the classroom can have both immediate and long-term impacts on their development. These interactions were highly associated with improvements in social skills, receptive language, expressive language, early literacy skills, and school preparation. Therefore, young children's health, growth, and learning are extremely dependent upon the mental health of their teachers, the quality of emotional support, and the positive responsive interactions between the teacher and the children.

For this reason, Arab Resource Collective (ARC) offers a Mental Health & Psychosocial Support (MHPSS) online toolkit tailored for ECD frontliners. Using a holistic and multidisciplinary approach, this toolkit will provide the adequate support, tools, and resources for ECD frontliners, which can improve their resilience and ability to cope with stressors, which in turn will promote their mental health and improve their job satisfaction and ultimately benefit the children they work with.

For the development of the MHPSS online toolkit, a needs assessment was conducted in partnership with Modern University for Business & Science (MUBS); a sample of 915 ECD frontliners answered an online questionnaire about mental health, psychological symptoms, coping skills, quality of life, work performance, and attitudes toward psychological interventions and emotional support. Based on this assessment (study), and based on the needs of ECD frontliners (as shown in the study results), the topics of the toolkit were identified.

The MHPSS online toolkit was developed by mental health experts and specialists using validated mental health resources; this toolkit is not a psychological therapy, it is a stress management toolkit, in which the techniques that were included were chosen carefully to help ECD frontliners deal with different stressors. It was also reviewed by mental health experts and education experts, and it was proofread in Arabic.

ELIGIBILITY:
Inclusion Criteria:

* ECD frontliners working directly with children under 8 years old in Lebanon (teachers, social workers, caretakers in nurseries, etc.).
* Individuals who are able to access and complete an online MHPSS toolkit.
* Individuals who are not currently employed in the mental health field.
* Participants who have not received prolonged mental health services (psychological therapy).

Exclusion Criteria:

* Professionals who work specifically in the mental health field (child psychologists, mental health support providers).
* Individuals who have received prolonged mental health services (to prevent potential bias due to prior mental health intervention experience).

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-01-20 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Change in psychological immunity among ECD Frontliners after participation in the web-based psychosocial support toolkit | Baseline (pre-intervention) to immediately post-intervention (after completion of the 10-session web-based toolkit; approximately 8 weeks).
  This outcome measures the change in participants' psychological immunity levels before and after completing the web-based psychosocial support toolkit. Psychological immunity reflects individuals' resilience, adaptability, regulation, and efficacy.
  The scale includes 40 items rated on a 5-point Likert scale (1 = strongly disagree to 5 = strongly agree) and comprises the following subscales: sense of control, creative self-concept, sense of self-growth, problem-solving capacity, self-efficacy, impulse control, emotional control, and irritability. Total scores range from 40 to 200, with higher scores indicating greater psychological immunity. Scores below 93 indicate low psychological immunity.
  The scale will be administered at baseline and immediately after completion of the web-based psychosocial support toolkit to assess changes associated with the intervention.
Change in cognitive emotional regulation among ECD Frontliners after participation in the web-based psychosocial support toolkit | Baseline (pre-intervention) to immediately post-intervention (after completion of the 10-session web-based toolkit; approximately 8 weeks)
  This outcome measures the change in participants' cognitive emotional regulation levels before and after completing the web-based psychosocial support toolkit.
  Cognitive emotion regulation will be assessed using the short Cognitive Emotion Regulation Questionnaire (CERQ), a self-report measure evaluating the cognitive strategies individuals use to manage emotional responses to stressful events. The questionnaire includes 18 items covering the following subscales: self-blame, acceptance, rumination, positive refocusing, refocus on planning, positive reappraisal, putting into perspective, catastrophizing, and other-blame.
  Items are rated on a Likert-type scale, yielding a total score ranging from 18 to 90, with higher scores indicating better cognitive emotion regulation abilities. Scores below 42 indicate low levels of cognitive emotion regulation.
Change in self-care behaviors among ECD Frontliners after participation in the web-based psychosocial support toolkit | Baseline (pre-intervention) to immediately post-intervention (after completion of the 10-session web-based psychosocial support toolkit; approximately 8 weeks)
  This outcome measures the change in participants' self-care behaviors levels before and after completing the web-based psychosocial support toolkit. Participants will complete a self-care behaviors scale at baseline (pre-test) and after completing the 10-session online intervention (post-test). Higher post-test scores will indicate improved self-care behaviors as a result of the intervention.
  Self-care behaviors will be assessed using the Mindful Self-Care Scale, a self-report instrument designed to evaluate individuals' engagement in mindful and supportive self-care practices. The scale includes 24 items across the following subscales: mindful relaxation, physical care, self-compassion and purpose, supportive relationships, supportive structure, and mindful awareness.
  Items are rated on a Likert-type scale, producing a total score ranging from 24 to 120, with higher scores indicating better self-care behaviors. Scores below 56 are considered indicative of low self-care behaviors.

SECONDARY OUTCOMES:
Change in job performance among ECD Frontliners after participation in the web-based psychosocial support toolkit | Baseline (pre-intervention) to immediately post-intervention (after completion of the 10-session web-based psychosocial support toolkit; approximately 8 weeks)
  This outcome measures the change in participants' job performance levels before and after completing the web-based psychosocial support toolkit. Participants will complete a job performance scale at baseline (pre-test) and after completing the 10-session online intervention (post-test). Higher post-test scores will indicate improved job performance as a result of the intervention.
  Job performance will be assessed using a Short Job Performance Scale, a self-report instrument designed to evaluate perceived work effectiveness, task completion, focus, and engagement in the workplace. The scale consists of 10 items rated on a Likert-type scale, yielding a total score ranging from 10 to 50.
  Higher scores indicate better job performance, while scores below 23 are considered indicative of low job performance.
  The scale will be administered at baseline and immediately after completion of the web-based psychosocial support toolkit to assess changes associated with the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Rasha Tadmori, Principal Investigator — Arab Resource Collective (ARC)
Locations (1):
- Arab Resource Collective, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No